CLINICAL TRIAL: NCT04998851
Title: A Phase IV Multicenter, Open-Label Study Evaluating B Cell Levels In Infants Of Lactating Women With CIS Or MS Receiving Ocrelizumab
Brief Title: A Study Evaluating B Cell Levels In Infants Of Lactating Women With CIS Or MS Receiving Ocrelizumab
Acronym: SOPRANINO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: PPD Development, LP (Industry); Laboratory Corporation of America (Industry); Illingworth Research Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MN42989; 2021-000063-79 (EudraCT Number)
Record Dates: First submitted 2021-08-06; First posted 2021-08-10 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: ocrelizumab, OCREVUS, breastmilk transfer, breast milk transfer, lactation
MeSH Terms: conditions — Multiple Sclerosis; Breast Feeding | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Women with CIS or MS (Experimental): Lactating women with CIS or MS (in line with the locally approved indications) who decided together with their treating physician to continue on, or start treatment with, OCREVUS (ocrelizumab) post-partum. Women resuming treatment with ocrelizumab post-partum will be included only if the last exposure to ocrelizumab occurred more than 3 months before the last menstrual period to exclude any interference between fetal exposure and exposure via lactation.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Women will receive the ocrelizumab dose regimen as per the locally-approved label. The ocrelizumab dose will be administered as an initial split dose of two 300 mg infusions separated by 14 days or a single 600 mg infusion according to the local prescribing information.

SUMMARY:
This study will evaluate the pharmacokinetics of ocrelizumab in the breastmilk of lactating women with clinically isolated syndrome (CIS) or multiple sclerosis (MS) [in line with the locally approved indications] treated with ocrelizumab, by assessing the concentration of ocrelizumab in mature breastmilk, as well as the corresponding exposure and pharmacodynamic effects (blood B cell levels) in the infants.

ELIGIBILITY:
Inclusion Criteria:

* Woman is between 18 and 40 years of age at screening
* Woman is willing to breastfeed for at least 60 days after the first post-partum ocrelizumab infusion (this decision is to be taken prior to and independent from study participation)
* Woman is willing to provide breastmilk samples
* Woman has a diagnosis of MS or CIS (in line with the locally approved indications)
* Woman has delivered a healthy term singleton infant (≥37 weeks gestation)
* Infant is between 2-24 weeks of age at the time of the mother's first post-partum dose of ocrelizumab
* For women who received commercial ocrelizumab (OCREVUS) before enrolment: documentation that last exposure to ocrelizumab occurred more than 3 months before the last menstrual period (LMP) and was given at the approved dose of 2 x 300 mg or 1 x 600 mg
* Woman agrees to use acceptable contraceptive methods during the study

Exclusion Criteria related to the Mother:

* Hypersensitivity to ocrelizumab or to any of its excipients
* Received last dose of ocrelizumab <3 months before the LMP or during pregnancy
* Active infections (may be included once the infection is treated and is resolved; women with bilateral mastitis infection should not have samples collected until the infection is completely resolved)
* Prior or current history of primary or secondary immunodeficiency, or woman in an otherwise severely immunocompromised state
* Known active malignancies, or being actively monitored for recurrence of malignancy
* History of breast implants, breast augmentation, breast reduction surgery or mastectomy
* Prior or current history of chronic alcohol abuse or drug abuse
* Positive screening tests for hepatitis B
* Treatment with a DMT for CIS or MS during pregnancy and/or first weeks post-partum, with the exception of formulations of interferon-beta, glatiramer acetate or pulsed corticosteroids
* Treatment with drugs known to transfer to the breastmilk and with established or potential deleterious effects for the infant
* Treatment with any investigational agent within 6 months or five half-lives of the investigational drug prior to the LMP

Exclusion Criteria related to the Infant:

* >24 weeks of life at the time of the mother's first dose of ocrelizumab
* Any abnormality that may interfere with breastfeeding or milk absorption
* Active infection (may be included once the infection resolves)
* Infant has any other medical condition or abnormality that, in the opinion of the investigator, could compromise the infant's ability to participate in this study, including interference with the interpretation of study results
* At least one documented brief resolved unexplained event (BRUE), as defined by the 2016 Guidelines of the American Academy of Pediatrics

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Lactating women with CIS or MS (in line with the locally approved indications) who decided together with their treating physician to continue on, or start treatment with, OCREVUS (ocrelizumab) post-partum. Women resuming treatment with ocrelizumab post-partum will be included only if the last exposure to ocrelizumab occurred more than 3 months before the last menstrual period to exclude any interference between fetal exposure and exposure via lactation.
Enrollment: 26 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Memorial Healthcare Institute for Neurosciences and Multiple Sclerosis, Owosso, Michigan
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Hosp. Clinico San Carlos, Madrid, Spain
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 mother-infant pairs took part in the study across 7 sites in the United States, Spain, and the United Kingdom from 16 September 2021 to 13 January 2025.
Pre-assignment Details: Lactating mothers with clinically isolated syndrome (CIS) or multiple sclerosis (MS) who, in consultation with their treating physician, chose to continue or start postpartum treatment with commercial ocrelizumab were enrolled in this study. This study included a 60-day treatment and sampling period followed by an 11-month vaccination period.
Groups:
- Mothers: Lactating mothers initiating ocrelizumab received two doses of 300 milligrams (mg), as an intravenous (IV) infusion on Day 1 and Day 14, and mothers resuming ocrelizumab received a single dose of 600 mg, as an IV infusion on Day 1 at the discretion of the physicians, in accordance with local prescribing information.
- Infants: Infants of mothers who received commercial IV ocrelizumab at the discretion of the physicians, in accordance with local prescribing information were observed until the last visit which was at 1 month (+ 30 days) after the first dose of measles, mumps, and rubella (MMR) vaccine (if first dose is administered at 11 months of age or later) or 1 month (+ 30 days) after second dose of MMR vaccine (if first dose is administered before 11 months of age), or at Month 13 of chronological age (+ 30 days) if MMR vaccine is not planned to be administered.
Period: Treatment and Sampling Period (60 Days)
Arm/Group | Mothers | Infants
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Vaccination Period (11 Months)
Arm/Group | Mothers | Infants
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set Mothers (SAFM) included all mothers who met the eligibility criteria and received any post-partum dose of ocrelizumab. Safety Analysis Set Infants (SAFI) included all the infants of women in the Full Analysis Set Mothers (FASM) population. As consent for race and ethnicity was not obtained, this data has not been reported.
Groups:
- Mothers: Lactating mothers initiating ocrelizumab received two doses of 300 mg, as an IV infusion on Day 1 and Day 14, and mothers resuming ocrelizumab received a single dose of 600 mg, as an IV infusion on Day 1 at the discretion of the physicians, in accordance with local prescribing information.
- Infants: Infants of mothers who received commercial IV ocrelizumab at the discretion of the physicians, in accordance with local prescribing information were observed until the last visit which was at 1 month (+ 30 days) after the first dose of MMR vaccine (if first dose is administered at 11 months of age or later) or 1 month (+ 30 days) after second dose of MMR vaccine (if first dose is administered before 11 months of age), or at Month 13 of chronological age (+ 30 days) if MMR vaccine is not planned to be administered.
- Total: Total of all reporting groups
Arm/Group | Mothers | Infants | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Customized [Count of Participants; unit: Participants]
  Preterm newborn infants (gestational age <37 weeks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 8 | 8
  Infants and toddlers (28 days-23 months) | 0 | 5 | 5
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 13 | 0 | 13
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 0 | 7 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not reported | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With B Cell Levels (Cluster of Differentiation 19 [CD19+] Cells) Below the Lower Limit of Normal (LLN) Measured at Day 30 After the Mother's First Ocrelizumab Postpartum Infusion
Description: Infant blood samples were collected at Day 30 after the mothers received their first postpartum ocrelizumab infusion (regardless of whether women receive a 600 mg or a 2x300 mg dose). The percentage of infants with B cell levels below LLN are reported with the two-sided Clopper Pearson 95% confidence interval (CI). B-cell reference ranges by week of life (absolute and percentage counts) are defined by Borriello et al. 2022.
Time Frame: At Day 30
Population: Full Analysis Set Infants (FASI) included all the infants of women in the FASM population. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 30.85]

2. Primary Outcome: Estimated Average Oral Daily Infant Dosage (ADID)
Description: ADID was calculated as the arithmetic mean of the mother's daily ocrelizumab milk concentration (micrograms/milliliters [µg/mL]) over 60 days post-ocrelizumab infusion 1 multiplied by an estimated infant milk intake of 150 milliliters/kilograms/day (mL/kg/day) and based on the weight [kilograms (kg)] recorded at the Day 30 visit. Ocrelizumab concentrations reported as below the lower limit of quantification [LLQ=160 nanograms/millilitres (ng/mL)] are imputed to zero for the calculation ADID.
Time Frame: Up to Day 60
Population: Pharmacokinetic Analysis Set Mothers (PASM) included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (95% Confidence Interval); unit: micrograms (µg)
Arm/Group | Mothers
Number analyzed (Participants) | 12
micrograms (µg) | 64.50 [21.415 to 107.587]

3. Secondary Outcome: Absolute CD19+ B Cell Count in the Infant
Description: Infant blood samples were collected at Day 30 after the mothers received their first postpartum ocrelizumab infusion (regardless of whether women receive a 600 mg or a 2x300 mg dose).
Time Frame: At Day 30
Population: FASI included all the infants of women in the FASM population. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: cells per microliter (cells/µL)
Arm/Group | Infants
Number analyzed (Participants) | 10
cells per microliter (cells/µL) | 1431.50 [869.0 to 2241.0]

4. Secondary Outcome: Percentage of CD19+ B Cell in the Infant
Description: as for outcome 3
Time Frame: At Day 30
Population: as for outcome 3
Measure: Median (Full Range); unit: percentage of cells
Arm/Group | Infants
Number analyzed (Participants) | 10
percentage of cells | 21.80 [10.0 to 31.7]

5. Secondary Outcome: Area Under the Milk Concentration-Time Curve (AUC) of Ocrelizumab in Mature Breastmilk
Time Frame: One 600 mg infusion: before infusion and at 24 hours (Day 1), Days 7, 30 and 60 post-infusion; Two 300 mg infusions: before infusion 1 and at 24 hours (Day 1), Days 7, 14, 15 (24 hours after infusion 2), 21, 30 and 60 post-infusion 1
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: micrograms/millilitres*day (μg/mL*day)
Arm/Group | Mothers
Number analyzed (Participants) | 12
micrograms/millilitres*day (μg/mL*day) | 3.98 (4.93)

6. Secondary Outcome: Average Concentration of Ocrelizumab in Breastmilk (Cmean)
Time Frame: as for outcome 5
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Mothers
Number analyzed (Participants) | 12
μg/mL | 0.074 (0.077)

7. Secondary Outcome: Maximum Concentration (Cmax) of Ocrelizumab in Breastmilk
Time Frame: as for outcome 5
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Mothers
Number analyzed (Participants) | 12
μg/mL | 0.18 (0.15)

8. Secondary Outcome: Time of Maximum Concentration (Tmax) of Ocrelizumab in Breastmilk
Time Frame: as for outcome 5
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Median (Full Range); unit: days
Arm/Group | Mothers
Number analyzed (Participants) | 12
days | 3.97 [0.00 to 59.9]

9. Secondary Outcome: Estimated Maximum Oral Daily Infant Dosage (MDID)
Description: MDID was calculated at the subject level as the peak ocrelizumab milk concentration (μg/mL) multiplied by an estimated infant milk intake of 150 mL/kg/day measured over 60 days after the mother's first postpartum ocrelizumab infusion.
Time Frame: Up to Day 60
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Mothers
Number analyzed (Participants) | 12
µg | 153.20 (137.15)

10. Secondary Outcome: Average Relative Infant Dose (RID)
Description: Average RID over 60 days was calculated as the ADID (mg/kg/day) divided by the maternal dosage (mg/kg/day) over 60 days multiplied by 100.
Time Frame: Up to Day 60
Population: PASM included all mothers in the FASM with a breastmilk sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Mothers
Number analyzed (Participants) | 12
percentage | 0.50 (0.58)

11. Secondary Outcome: Serum Concentration of Ocrelizumab in the Infant at Day 30
Description: Serum concentration of ocrelizumab in the infant measured at Day 30 after the mother's first ocrelizumab postpartum infusion. Concentrations reported as below the lower limit of quantification (LLQ=156 ng/mL) are set to zero for calculation of summary statistics.
Time Frame: At Day 30
Population: Pharmacokinetic Analysis Set Infants (PASI) included all infants in the FASI with a serum sample to allow measurement of ocrelizumab concentration.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Infants
Number analyzed (Participants) | 9
µg/mL | NA (NA) — Mean and standard deviation was not evaluable as the samples were below the limit of quantification (BLQ).

12. Secondary Outcome: Percentage of Mothers With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: Up to approximately 73.3 weeks after first ocrelizumab dose
Population: Safety Analysis Set Mothers (SAFM) included all mothers who met the eligibility criteria and received any post-partum dose of ocrelizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Mothers
Number analyzed (Participants) | 13
percentage of participants | 76.9

13. Secondary Outcome: Percentage of Infants With AEs
Description: as for outcome 12
Time Frame: Up to approximately 73.3 weeks after first ocrelizumab dose administered to mother
Population: Safety Analysis Set Infants (SAFI) included all the infants of women in the FASM population.
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 13
percentage of infants | 92.3

14. Secondary Outcome: Mean Titers of Measles, Immunoglobin G (IgG) Antibody in Response to Measles, Mumps, and Rubella (MMR) Vaccination
Description: The immune response to MMR vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines. mIU/mL=milli-international units per milliliter.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: Antibody Immune Response Analysis Set of Infants (AIRI) included all infants in the SAFI for whom any serum titers of antibody immune response to vaccinations were available.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Infants
Number analyzed (Participants) | 11
mIU/mL | 2590.91 (2210.74)

15. Secondary Outcome: Mean Titers of Mumps, IgG Antibody in Response to MMR Vaccination
Description: The immune response to MMR vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines. RU/mL=relative units per milliliter.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: AIRI included all infants in the SAFI for whom any serum titers of antibody immune response to vaccinations were available. Overall number analyzed are the number of infants with data available for analysis.
Measure: Mean (Standard Deviation); unit: RU/mL
Arm/Group | Infants
Number analyzed (Participants) | 9
RU/mL | 54.19 (34.72)

16. Secondary Outcome: Mean Titers of Rubella, IgG Antibody in Response to MMR Vaccination
Description: The immune response to MMR vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines. IU/mL=international units per milliliter.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Infants
Number analyzed (Participants) | 10
IU/mL | 94.21 (51.39)

17. Secondary Outcome: Percentage of Infants With Positive Humoral Response to MMR Vaccination
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) was presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for MMR vaccine are as follows: Anti-Measles Vir IgG(-70)CL: ≥ 120 mIU/mL; Anti-MumpsAT Vir iGG(-70)CL: ≥ 17 RU/mL; Anti-Rub Vir IgG(-70)RUOCL: ≥ 10 IU/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: AIRI included all infants in the SAFI for whom any serum titers of antibody immune response to vaccinations were available. Number analyzed refers to infants with data available for the specified IgG antibody titer.
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 11
percentage of infants
  Measles, IgG | 100
  Mumps, IgG: number analyzed (Participants) | 9
  Mumps, IgG | 77.8
  Rubella, IgG: number analyzed (Participants) | 10
  Rubella, IgG | 100

18. Secondary Outcome: Mean Titers of Corynebacterium Diphtheriae, IgG Antibody in Response to Diphtheria-Tetanus-Pertussis (DTP) Vaccine
Description: The immune response to DTP vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Infants
Number analyzed (Participants) | 10
IU/mL | 1.94 (3.13)

19. Secondary Outcome: Mean Titers of Bordetella Pertussis, IgG Antibody in Response to DTP Vaccine
Description: The immune response to DTP vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. Cut-off Index (COI) = unitless ratio calculated as the signal intensity of the sample divided by the signal of the assay's cut-off calibrator. It is interpreted as follows:
  * COI < 0.95: Negative
  * COI 0.95-1.04: Equivocal
  * COI > 1.04: Positive The assay used has not been standardized against WHO International Units (IU/mL) for Bordetella pertussis IgG and therefore, cannot be converted to IU/mL. Higher COI values = a stronger antibody signal, but are not directly correlated with clinical protection. Positivity was defined using the manufacturer's COI cut-off (>1.04).
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: COI
Arm/Group | Infants
Number analyzed (Participants) | 10
COI | 1.12 (0.82)

20. Secondary Outcome: Mean Titers of Tetanus Toxoid, IgG Antibody in Response to DTP Vaccine
Description: as for outcome 18
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Infants
Number analyzed (Participants) | 6
IU/mL | 1.23 (0.43)

21. Secondary Outcome: Percentage of Infants With Positive Humoral Response to DTP Vaccine
Description: as for outcome 19
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: AIRI included all infants in the SAFI for whom any serum titers of antibody immune response to vaccinations were available. Overall number analyzed are the number of infants with data available for analysis. Number analyzed refers to infants with data available for the specified IgG antibody titer.
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 10
percentage of infants
  Corynebacterium Diphtheriae, IgG | 100
  Bordetella Pertussis, IgG | 50
  Tetanus Toxoid, IgG: number analyzed (Participants) | 6
  Tetanus Toxoid, IgG | 100

22. Secondary Outcome: Mean Titers of Haemophilus Influenzae Type B (Hib), IgG Antibody in Response to Hib Vaccine
Description: The immune response to Hib vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Infants
Number analyzed (Participants) | 9
micrograms per milliliter (ug/mL) | 3.45 (4.21)

23. Secondary Outcome: Percentage of Infants With Positive Humoral Response to Hib Vaccine
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) was presented for the IgG antibody titer. Seroprotective titer based on vaccine tests for Hib vaccine are as follows: Hib, IgG: ≥ 0.15 µg/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 9
percentage of infants | 88.9

24. Secondary Outcome: Mean Titers of Anti-Hepatitis B Surface Antibody in Response to Hepatitis B Virus (HBV) Vaccine
Description: The immune response to HBV vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Infants
Number analyzed (Participants) | 7
mIU/mL | 1158.01 (1263.32)

25. Secondary Outcome: Percentage of Infants With Positive Humoral Response to HBV Vaccine
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) was presented for the IgG antibody titer. Seroprotective titer based on vaccine tests for HBV vaccine are as follows: Anti-HBs: ≥ 10 mIU/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 7
percentage of infants | 100

26. Secondary Outcome: Mean Titers of Pneumococcal Capsular Polysaccharide, Serotypes, IgG Antibody in Response to 13-valent Pneumococcal Conjugate Vaccine (PCV-13)
Description: The immune response to PCV-13 vaccine was assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine was not planned to be administered. This was to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Infants
Number analyzed (Participants) | 10
ug/mL
  Pneumococcal Capsular Polysaccharide, Serotype 1, IgG | 4.80 (6.38)
  Pneumococcal Capsular Polysaccharide, Serotype 3, IgG | 2.56 (3.16)
  Pneumococcal Capsular Polysaccharide, Serotype 4, IgG | 8.28 (9.18)
  Pneumococcal Capsular Polysaccharide, Serotype 5, IgG | 9.98 (15.72)
  Pneumococcal Capsular Polysaccharide, Serotype 6A, IgG | 27.28 (34.50)
  Pneumococcal Capsular Polysaccharide, Serotype 6B, IgG | 27.02 (70.85)
  Pneumococcal Capsular Polysaccharide, Serotype 7F, IgG | 9.44 (14.11)
  Pneumococcal Capsular Polysaccharide, Serotype 9V, IgG | 4.21 (3.66)
  Pneumococcal Capsular Polysaccharide, Serotype 14, IgG | 14.93 (14.49)
  Pneumococcal Capsular Polysaccharide, Serotype 18C, IgG | 9.62 (11.47)
  Pneumococcal Capsular Polysaccharide, Serotype 19A, IgG | 1.70 (1.41)
  Pneumococcal Capsular Polysaccharide, Serotype 19F, IgG | 45.83 (80.11)
  Pneumococcal Capsular Polysaccharide, Serotype 23F, IgG | 10.50 (13.17)

27. Secondary Outcome: Percentage of Infants With Positive Humoral Response to PCV-13
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) was presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for PCV-13 vaccine are as follows: 13 Valent anti-pneumococcal antibody panel: ≥ 0.35 µg/ml.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Population: as for outcome 15
Measure: Number; unit: percentage of infants
Arm/Group | Infants
Number analyzed (Participants) | 10
percentage of infants
  Pneumococcal Capsular Polysaccharide, Serotype 1, IgG | 80
  Pneumococcal Capsular Polysaccharide, Serotype 3, IgG | 70
  Pneumococcal Capsular Polysaccharide, Serotype 4, IgG | 80
  Pneumococcal Capsular Polysaccharide, Serotype 5, IgG | 90
  Pneumococcal Capsular Polysaccharide, Serotype 6A, IgG | 100
  Pneumococcal Capsular Polysaccharide, Serotype 6B, IgG | 80
  Pneumococcal Capsular Polysaccharide, Serotype 7F, IgG | 100
  Pneumococcal Capsular Polysaccharide, Serotype 9V, IgG | 90
  Pneumococcal Capsular Polysaccharide, Serotype 14, IgG | 100
  Pneumococcal Capsular Polysaccharide, Serotype 18C, IgG | 80
  Pneumococcal Capsular Polysaccharide, Serotype 19A, IgG | 60
  Pneumococcal Capsular Polysaccharide, Serotype 19F, IgG | 100
  Pneumococcal Capsular Polysaccharide, Serotype 23F, IgG | 80

ADVERSE EVENTS:
Time Frame: Mothers and Infants: Up to approximately 73.3 weeks
Description: SAFM included all mothers who met the eligibility criteria and received any post-partum dose of ocrelizumab. SAFI included all the infants of women in the FASM population.
Arm/Group | Mothers | Infants
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 10/13 | 12/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mothers (N=13) | Infants (N=13)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (2)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 4 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 3 (4)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis pseudo relapse (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (2) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04998851/Prot_002.pdf
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04998851/SAP_001.pdf